CLINICAL TRIAL: NCT05826210
Title: Effect of Sarcopenic Obesity on Weight Loss Outcomes and Quality of Life After Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Prof., Fujian Medical University Union Hospital
Other Study IDs: 2023-03
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenic Obesity; Body Composition
Keywords: laparoscopic sleeve gastrectomy; weight loss; sarcopenic obesity; Fat-free mass; Quality of life
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenic obesity group: Patients who underwent LSG with FM/FFM>0.80 calculated from the cross-sectional CT image of L3 vertebra.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Non-sarcopenic obesity group: Patients who underwent LSG with FM/FFM<0.80 calculated from the cross-sectional CT image of L3 vertebra.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic sleeve gastrectomy was performed in all patients with or without SO.

SUMMARY:
The purpose of this study is to assess the impact of sarcopenic obesity (SO) on weight loss outcomes and improvement of quality of life after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Sarcopenic obesity is a state in which a lack of muscle mass and strength coexists with an increase in fat mass, and it may affect the health outcome of people with obesity after laparoscopic sleeve gastrectomy (LSG).No studies have reported differences in weight loss outcomes between patients with SO and those with non-sarcopenic obesity (NSO) after LSG. Therefore, this study aimed to systematically evaluate the differences in weight loss and quality of life (QOL) evaluation between patients with SO and NSO after LSG and provide high-level evidence-based medical evidence for the impact of SO on weight loss in the obese population and refinement of follow-up strategies.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients who met the indications for LSG and were followed up regularly as planned after surgery.

Exclusion Criteria:

1. incomplete critical clinical data;
2. incomplete imaging data;
3. insufficient follow-up data.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective monocentric study included 260 obese patients who underwent LSG between January 2015 and July 2022 at the Department of Gastric Surgery, Fujian Medical University Union Hospital. All patients underwent a thorough multidisciplinary evaluation (an endocrinologist, dietician, and bariatric surgeon), and a psychiatric evaluation was obtained if considered necessary. All patients completed routine preoperative investigations, including upper gastrointestinal endoscopy, chest radiography, abdominal computed tomography (CT), abdominal ultrasound examination, and nutritional assessment. Preoperative QOL was measured using the Moorhead-Ardelt questionnaire at the same visit.
  All patients in this study were operated on by the same surgical team of surgeons with more than 60 LSG experiences.Postoperative treatment was performed based on the patient's condition.
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
%EWL | 6 month after surgery
  Percentage excess weight loss is calculated as (initial weight - 6-month weight)/(initial weight - ideal weight) × 100%.

SECONDARY OUTCOMES:
%EWL | 1 month after surgery
  Percentage excess weight loss is calculated as (initial weight - 1-month weight)/(initial weight - ideal weight) × 100%.
%EWL | 3 month after surgery
  Percentage excess weight loss is calculated as (initial weight - 3-month weight)/(initial weight - ideal weight) × 100%.
%EWL | 9 month after surgery
  Percentage excess weight loss is calculated as (initial weight - 9-month weight)/(initial weight - ideal weight) × 100%.
%EWL | 12 month after surgery
  Percentage excess weight loss is calculated as (initial weight - 12-month weight)/(initial weight - ideal weight) × 100%.
%TWL | 6 month after surgery
  Percentage total weight loss is calculated as (initial weight - 6-month weight)/(initial weight) × 100%
%TWL | 12 month after surgery
  Percentage total weight loss is calculated as (initial weight - 12-month weight)/(initial weight) × 100%
EBMI | 6 month after surgery
  Excess BMI is calculated as(follow-up BMI - ideal BMI)
%WL | 6 month after surgery
  Percentage weight loss is calculated as (follow-up weight/initial weight) × 100%
MA II score | 6 month after surgery
  Moorhead-Ardelt QOL questionnaire is a six-item self-report questionnaire that assesses the patient's subjective impression of QOL,The total score ranges from -3 to +3 and defines five outcome groups: very poor, poor, fair, good, and very good. Good and very good outcomes were considered satisfactory.
BAROS score | 6 month after surgery
  The Bariatric Analysis and Reporting Outcome System(BAROS)combines the Moorhead-Ardelt QOL questionnaire with other data relevant to bariatric surgery, including the %EWL, improvement in comorbid conditions, and complications.A BAROS score ≤1 was considered a failure; >1-3, fair; >3-5, good; >5-7, very good; and >7, excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Ph.D, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Chang-ming Huang, Fuzhou, Fujian, China

REFERENCES:
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Sung H, Siegel RL, Torre LA, Pearson-Stuttard J, Islami F, Fedewa SA, Goding Sauer A, Shuval K, Gapstur SM, Jacobs EJ, Giovannucci EL, Jemal A. Global patterns in excess body weight and the associated cancer burden. CA Cancer J Clin. 2019 Mar;69(2):88-112. doi: 10.3322/caac.21499. Epub 2018 Dec 12. PMID 30548482
- [Background] Panagiotou OA, Markozannes G, Adam GP, Kowalski R, Gazula A, Di M, Bond DS, Ryder BA, Trikalinos TA. Comparative Effectiveness and Safety of Bariatric Procedures in Medicare-Eligible Patients: A Systematic Review. JAMA Surg. 2018 Nov 1;153(11):e183326. doi: 10.1001/jamasurg.2018.3326. Epub 2018 Nov 21. PMID 30193303
- [Background] Thibault R, Genton L, Pichard C. Body composition: why, when and for who? Clin Nutr. 2012 Aug;31(4):435-47. doi: 10.1016/j.clnu.2011.12.011. Epub 2012 Jan 31. PMID 22296871
- [Background] Prado CM, Wells JC, Smith SR, Stephan BC, Siervo M. Sarcopenic obesity: A Critical appraisal of the current evidence. Clin Nutr. 2012 Oct;31(5):583-601. doi: 10.1016/j.clnu.2012.06.010. Epub 2012 Jul 17. PMID 22809635
- [Background] Kim TN, Choi KM. Sarcopenia: definition, epidemiology, and pathophysiology. J Bone Metab. 2013 May;20(1):1-10. doi: 10.11005/jbm.2013.20.1.1. Epub 2013 May 13. PMID 24524049
- [Background] Dhana K, Koolhaas CM, Schoufour JD, Rivadeneira F, Hofman A, Kavousi M, Franco OH. Association of anthropometric measures with fat and fat-free mass in the elderly: The Rotterdam study. Maturitas. 2016 Jun;88:96-100. doi: 10.1016/j.maturitas.2016.03.018. Epub 2016 Apr 1. PMID 27105706
- [Background] Low S, Goh KS, Ng TP, Ang SF, Moh A, Wang J, Ang K, Subramaniam T, Sum CF, Lim SC. The prevalence of sarcopenic obesity and its association with cognitive performance in type 2 diabetes in Singapore. Clin Nutr. 2020 Jul;39(7):2274-2281. doi: 10.1016/j.clnu.2019.10.019. Epub 2019 Nov 4. PMID 31744622
- [Background] Baracos VE, Arribas L. Sarcopenic obesity: hidden muscle wasting and its impact for survival and complications of cancer therapy. Ann Oncol. 2018 Feb 1;29(suppl_2):ii1-ii9. doi: 10.1093/annonc/mdx810. PMID 29506228
- [Background] Hong SH, Choi KM. Sarcopenic Obesity, Insulin Resistance, and Their Implications in Cardiovascular and Metabolic Consequences. Int J Mol Sci. 2020 Jan 13;21(2):494. doi: 10.3390/ijms21020494. PMID 31941015
- [Background] Huang R, Gagner M. A Thickness Calibration Device Is Needed to Determine Staple Height and Avoid Leaks in Laparoscopic Sleeve Gastrectomy. Obes Surg. 2015 Dec;25(12):2360-7. doi: 10.1007/s11695-015-1705-8. PMID 26024735
- [Background] Xu G, Song M. Recent advances in the mechanisms underlying the beneficial effects of bariatric and metabolic surgery. Surg Obes Relat Dis. 2021 Jan;17(1):231-238. doi: 10.1016/j.soard.2020.08.028. Epub 2020 Aug 31. PMID 33036939
- [Background] Manoy P, Anomasiri W, Yuktanandana P, Tanavalee A, Ngarmukos S, Tanpowpong T, Honsawek S. Elevated serum leptin levels are associated with low vitamin D, sarcopenic obesity, poor muscle strength, and physical performance in knee osteoarthritis. Biomarkers. 2017 Dec;22(8):723-730. doi: 10.1080/1354750X.2017.1315615. Epub 2017 Apr 19. PMID 28374624
- [Background] Shetty GK, Matarese G, Magkos F, Moon HS, Liu X, Brennan AM, Mylvaganam G, Sykoutri D, Depaoli AM, Mantzoros CS. Leptin administration to overweight and obese subjects for 6 months increases free leptin concentrations but does not alter circulating hormones of the thyroid and IGF axes during weight loss induced by a mild hypocaloric diet. Eur J Endocrinol. 2011 Aug;165(2):249-54. doi: 10.1530/EJE-11-0252. Epub 2011 May 20. PMID 21602313
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542